CLINICAL TRIAL: NCT03362879
Title: COSMOS - COmedication Study Assessing Mono- and cOmbination Therapy With Levodopa-carbidopa inteStinal Gel
Brief Title: COmedication Study Assessing Mono- and cOmbination Therapy With Levodopa-carbidopa inteStinal Gel
Acronym: COSMOS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-831
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: Advanced Parkinson's Disease; Levodopa-Carbidopa Intestinal Gel (LCIG)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with advanced Parkinson's disease: Participants with advanced Parkinson's disease on current treatment with levodopa-carbidopa intestinal gel (LCIG) for at least 12 months.

SUMMARY:
The purpose of this study is to evaluate treatment of advanced Parkinson's Disease (PD) patients on levodopa-carbidopa intestinal gel (LCIG) monotherapy in a routine clinical setting.

DETAILED DESCRIPTION:
Participants with advanced Parkinson's Disease who have been prescribed LCIG for at least 12 months will be entered into the study cohort. Clinical data will be collected by retrospective review of the participant's medical records as well as a single study visit for current data. Treatment of the participants and follow up will be according to the physician's judgment, regional regulations and the product monograph.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with APD and on LCIG treatment for at least 12 months
* Participant must have been on continuous LCIG treatment for at least 80% of days in the preceding year
* Participants must be treated by the same physician (principal investigator or co-investigator) since the initiation of LCIG treatment

Exclusion Criteria:

* Participation in a concurrent or a previous interventional clinical trial during which the participant was on LCIG therapy
* Lack of motivation or insufficient language skills to complete the study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with advanced Parkinson's disease (APD), on current treatment with levodopa-carbidopa intestinal gel (LCIG), and treated with LCIG for at least 12 months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (30):
- Austria (2):
  - Gailtal Klinik /ID# 202505, Hermagor-Pressegger See, Carinthia
  - Medizinische Universität Graz /ID# 202559, Graz, Styria
- Canada (4):
  - University of Calgary /ID# 206550, Calgary, Alberta
  - Ottawa Hospital /ID# 169448, Ottawa, Ontario
  - Toronto Western Hospital /ID# 169038, Toronto, Ontario
  - Clinique Neuro Levis /ID# 206549, Lévis, Quebec
- Clinical Hosp Center Zagreb /ID# 203553, Zagreb, Croatia
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne /ID# 209774, Brno, Brno-mesto
  - Fakultni Nemocnice Olomouc /ID# 209776, Olomouc, Olomoucký kraj
  - Vseobecna Fakultni Nemocnice /ID# 209775, Prague
- Greece (4):
  - Aiginiteio University Hospital /ID# 203476, Athens, Attica
  - HYGEIA Hospital /ID# 203474, Athens
  - Mediterraneo Hospital /ID# 203472, Glyfada
  - University Hospital of Ioannin /ID# 203471, Ioannina
- Hungary (4):
  - Pecsi Tudomanyegyetem /ID# 170026, Pécs, Pecs
  - Semmelweis Egyetem /ID# 170025, Budapest
  - Borsod-Abauj-Zemplen Megyei /ID# 170027, Miskolc
  - Szegedi Tudomanyegyetem /ID# 170028, Szeged
- Ireland (2):
  - Bon Secours Hospital /ID# 168424, Cork
  - University Hospital Galway /ID# 170754, Galway
- Israel (2):
  - Tel Aviv Sourasky Medical Ctr /ID# 167542, Tel Aviv, Tel Aviv
  - Sheba Medical Center /ID# 167543, Ramat Gan
- Romania (5):
  - Clinic Fundeni Institute /ID# 169265, Bucharest, București
  - Colentina Clinical Hospital /ID# 169263, Bucharest
  - Emergency Clinical County Hosp /ID# 169269, Târgu Mureş
  - Timisoara County /ID# 169266, Timișoara
  - Timisoara County /ID# 169268, Timișoara
- AbbVie Farmaceutica SLU /ID# 164364, Madrid, Spain
- Sweden (2):
  - Centrum for neurologi /ID# 171391, Stockholm
  - Neurologmottagningen /ID# 171390, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fasano A, Garcia-Ramos R, Gurevich T, Jech R, Bergmann L, Sanchez-Solino O, Parra JC, Simu M. Levodopa-carbidopa intestinal gel in advanced Parkinson's disease: long-term results from COSMOS. J Neurol. 2023 May;270(5):2765-2775. doi: 10.1007/s00415-023-11615-3. Epub 2023 Feb 18. PMID 36802031
- [Derived] Kovacs N, Szasz J, Vela-Desojo L, Svenningsson P, Femia S, Parra JC, Sanchez-Solino O, Bergmann L, Gurevich T, Fasano A. Motor and nonmotor symptoms in patients treated with 24-hour daily levodopa-carbidopa intestinal gel infusion: Analysis of the COmedication Study assessing Mono- and cOmbination therapy with levodopa-carbidopa inteStinal gel (COSMOS). Parkinsonism Relat Disord. 2022 Dec;105:139-144. doi: 10.1016/j.parkreldis.2022.08.002. Epub 2022 Aug 17. PMID 36008198
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 412 participants were enrolled in the study and 409 of these participants fulfilled all inclusion and none of the exclusion criteria and, thus, were included in the full analysis set.
Period: Overall Study
Arm/Group | Participants With Advanced Parkinson's Disease
Started | 409
Completed | 409
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the full analysis set (FAS) population (409) vs. enrolled (412).
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 405
  Asian | 2
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Levodopa-Carbidopa Intestinal Gel (LCIG) Monotherapy From LCIG Initiation to 12 Months
Description: The percentage of participants on LCIG monotherapy from immediately following LCIG initiation to 12 months. LCIG monotherapy means that the participant is not on any add-on Parkinson's (PD) medication/PD therapy at the respective time point (monotherapy 1) or that the participant is allowed to take an add-on PD medication/PD therapy at the respective time point but only in the evening after the LCIG infusion is completed (monotherapy 2).
Time Frame: 12 months
Population: Full analysis set (FAS): Participants that fulfilled all inclusion and none of the exclusion criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
percentage of participants
  Monotherapy 1 | 29.3
  Monotherapy 2 | 52.3

2. Secondary Outcome: Percentage of Participants Starting Add-On PD Medication Within 12 Months of LCIG Monotherapy Initiation
Description: LCIG monotherapy means that the participant is not on any add-on PD medication/PD therapy at the respective time point (monotherapy 1) or that the participant is allowed to take an add-on PD medication/PD therapy at the respective time point but only in the evening after the LCIG infusion is completed (monotherapy 2). PD medications were captured by time point and category from the initiation of LCIG therapy until the introduction of each add-on PD medication taken. Categories included levodopa, catechol-O-methyltransferase (COMT) inhibitors,dopamine agonist (excluding apomorphine), monoamine oxidase (MAO) inhibitor, n-methyl-d-aspartate receptor (NMDA) antagonist, apomorphine, anticholinergics, surgical therapy, or other. Participants may have initiated more than one PD medication or category.
Time Frame: 12 months
Population: FAS of participants starting add-on medication
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 260
percentage of participants
  Levodopa/carbidopa | 35.0
  Levodopa/benserazide | 23.8
  Levodopa/carbidopa/entacapone | 7.3
  Pramipexole | 15.4
  Rotigotine | 13.8
  Ropinirole | 11.5
  Rasagiline | 15.4
  Safinamide | 0.8
  Selegiline | 0.8
  Amantadine | 16.9
  Other | 5.0
  Anticholinergics | 2.7
  Deep brain stimulation | 1.2
  Pallidotomy | 0.4
  Entacapone | 1.2

3. Secondary Outcome: Total Daily Dose (in Milliliters) of LCIG Infusion at 12 Months After LCIG Initiation
Description: Physicians were asked to document the LCIG infusion details at 12 months after LCIG initiation, including the total daily dose. Total dose per day was calculated as morning dose + continuous dose x duration of infusion + extra dose. Abbreviations: ml = milliliters.
Time Frame: 12 months
Population: FAS and only participants with non-missing data.
Measure: Mean (Standard Deviation); unit: total LCIG dose per day (ml)
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 377
total LCIG dose per day (ml) | 69.2 (26.0)

4. Secondary Outcome: Healthcare Resource Utilization (HCRU): Primary Occupation by Number of Participants
Description: The HCRU questionnaire is used to assess healthcare resource utilization. Participants were asked about their occupational status (primary occupation), caregiver support (change in amount of caregiver help needed with daily activities/home care), and participant´s opinion on Parkinson's disease medication (number of pills in addition to LCIG the participant was willing to take each day).
  Physicians were asked to report details regarding participant visits and hospital admissions in the 12 months prior to the study visit.
Time Frame: 12 months
Population: FAS
Measure: Number; unit: participants
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
participants
  Retired | 372
  On sick leave | 6
  Unemployed | 16
  Working full time | 5
  Working part-time | 10

5. Secondary Outcome: HCRU: Caregiver Support by Number of Participants
Description: as for outcome 4
Time Frame: 12 months
Population: FAS
Measure: Number; unit: participants
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
participants
  Less help with daily activities or home care | 160
  More help with daily activities or home care | 83
  About same amount help daily activities/home care | 96
  Patient does not remember | 5
  Patient does not require any help | 65

6. Secondary Outcome: Percentage of Physicians With Overall Preference for LCIG Monotherapy
Description: The overall preference for treatment using LCIG as monotherapy compared with LCIG plus add-on PD medication, as stated by the physician.
Time Frame: 12 months
Population: Number of physicians stating LCIG as monotherapy is their overall treatment preference.
Measure: Number; unit: percentage of physicians
Groups:
- Percentage of Physicians: Percentage of Physicians with Overall Preference for LCGI Monotherapy.
Arm/Group | Percentage of Physicians
Number analyzed (Participants) | 56
percentage of physicians
  LCIG as monotherapy | 71.4
  LCIG plus add-on PD medication | 28.6

7. Secondary Outcome: Predictors for Monotherapy (Participant Data): Forward Selection for Monotherapy 1 (12 Months After LCIG Initiation)
Description: LCIG monotherapy 1 means that the participant is not on any add-on Parkinson's (PD) medication/PD therapy at the respective time point. The influence of predefined variables was evaluated using multivariable logistic regression models. The target variables were analyzed using two different sets of potential predictors: one set containing participant data and one set containing site and physician data.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: odds ratio estimate
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
odds ratio estimate
  Number of motor symptoms | 0.842 [0.751 to 0.944]
  Any dopamine agonists in the past Yes | 1.564 [0.999 to 2.450]
  Gross National Income | 0.974 [0.957 to 0.991]

8. Secondary Outcome: Predictors for Monotherapy (Physician Data): Forward Selection for Monotherapy 1 (12 Months After LCIG Initiation)
Description: LCIG monotherapy 1 means that the participant is not on any add-on Parkinson's (PD) medication/PD therapy at the respective time point. The influence of predefined variables was evaluated using multivariable logistic regression models. The target variables were analyzed using two different sets of potential predictors: one set containing participant data and one set containing site and physician data.
  Physician data in table shown as "average frequency of routine visits" includes average frequency of routine visits for advanced Parkinson's disease (APD) participants on device aided therapy ≥3x/years.
Time Frame: 12 months
Population: FAS
Measure: Number (95% Confidence Interval); unit: odds ratio estimate
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
odds ratio estimate
  Average frequency of routine visits | 2.760 [1.504 to 5.066]
  Average number of PD and APD participants per year | 1.000 [0.999 to 1.000]

9. Secondary Outcome: Duration (Days) of LCIG Monotherapy 1 or Monotherapy 2
Description: LCIG monotherapy means that the participant is not on any add-on PD medication/PD therapy at the respective time point (monotherapy 1) or that the participant is allowed to take an add-on PD medication/PD therapy at the respective time point but only in the evening after the LCIG infusion is completed (monotherapy 2). Duration of LCIG monotherapy was calculated for all participants who reached the respective monotherapy as time from LCIG initiation until LCIG is given as a monotherapy (separately for monotherapy 1 and monotherapy 2 definition).
Time Frame: 12 months
Population: FAS participants who reached the respective monotherapy (monotherapy 1 or monotherapy 2)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
days
  Duration of LCIG monotherapy 1 | 932.6 (621.5)
  Duration of LCIG monotherapy 2 | 945.1 (645.7)

10. Secondary Outcome: Time (Days) From Initial LCIG Administration to Substantial Dose Adjustments by Country
Description: Time for substantial change was determined as the time from LCIG initiation until the first substantial dose change in days 12 months after LCIG initiation. A substantial change was defined as a change of at least 20% compared to the LCIG dose at LCIG initiation.
Time Frame: 12 months
Population: FAS that includes only participants with substantial dose adjustments by each country that had participants meeting these criteria
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
days
  Austria: number analyzed (Participants) | 7
  Austria | 111.7 (80.6)
  Canada: number analyzed (Participants) | 9
  Canada | 283.2 (181.0)
  Czech Republic: number analyzed (Participants) | 17
  Czech Republic | 298.9 (770.1)
  Hungary: number analyzed (Participants) | 14
  Hungary | 387.4 (446.7)
  Israel: number analyzed (Participants) | 12
  Israel | 343.2 (423.7)
  Romania: number analyzed (Participants) | 10
  Romania | 460.8 (501.8)
  Spain: number analyzed (Participants) | 18
  Spain | 534.9 (750.1)
  Sweden: number analyzed (Participants) | 9
  Sweden | 394.7 (463.5)

11. Secondary Outcome: Time (Days) From Initial LCIG Administration to Substantial Dose Adjustment
Description: as for outcome 10
Time Frame: 12 months
Population: FAS that includes only participants with substantial dose adjustments
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 122
days | 409.2 (555.5)

12. Secondary Outcome: Days From Initial LCIG Administration to the Initiation of LCIG Monotherapy
Description: Time (in days) from LCIG initiation until monotherapy was calculated for those participants who were not on monotherapy (i.e., needed additional PD medication during LCIG infusion) at LCIG initiation, but reached monotherapy during the study. LCIG monotherapy means that the participant is not on any add-on PD medication/PD therapy at the respective time point (monotherapy 1) or that the participant is allowed to take an add-on PD medication/PD therapy at the respective time point but only in the evening after the LCIG infusion is completed (monotherapy 2).
Time Frame: 12 months
Population: FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
days
  Until Monotherapy 1 | 89.5 (220.9)
  Until Monotherapy 2 | 70.4 (240.1)

13. Secondary Outcome: Tapering Duration (Days) From Initial LCIG Administration of Each PD Medication
Description: LCIG monotherapy means that the participant is not on any add-on PD medication/PD therapy at the respective time point (monotherapy 1). The number of days for tapering process is the number of days between maximum and minimum daily dose; participants with minimum (or maximum, respectively) daily dose not at the end of the tapering process were checked. A maximum duration of approximately 2 months of the tapering process was allowed (otherwise the tapering process was set to missing).
Time Frame: 12 months
Population: FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Participants With Advanced Parkinson's Disease
Number analyzed (Participants) | 409
days
  Levodopa/carbidopa: number analyzed (Participants) | 5
  Levodopa/carbidopa | 21.3 (13.6)
  Levodopa/benserazide: number analyzed (Participants) | 2
  Levodopa/benserazide | 34.0 (11.3)
  Levodopa/carbidopa/entacapone: number analyzed (Participants) | 6
  Levodopa/carbidopa/entacapone | 21.0 (17.5)
  Entacapone: number analyzed (Participants) | 3
  Entacapone | 9.0 (7.0)
  Pramipexole: number analyzed (Participants) | 3
  Pramipexole | 34.3 (26.5)
  Ropinirole: number analyzed (Participants) | 2
  Ropinirole | 24.0 (2.8)
  Rotigotine: number analyzed (Participants) | 1
  Rotigotine | 6.0 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.
  Safinamide: number analyzed (Participants) | 1
  Safinamide | 32.0 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.
  Rasagiline: number analyzed (Participants) | 1
  Rasagiline | 57.0 (NA) — Standard deviation not calculated due to insufficient number of participants analyzed.
  Amantadine: number analyzed (Participants) | 3
  Amantadine | 34.3 (25.1)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Participants With Advanced Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/409
Serious Adverse Events (participants affected / at risk) | 0/409
Other Adverse Events (participants affected / at risk) | 0/409

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03362879/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT03362879/SAP_001.pdf